CLINICAL TRIAL: NCT03266224
Title: Digital Analysis of Ultrasonographic Images in Children With Wry Neck
Status: Completed | Type: Observational
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Chu-Hsu Lin, Principal Investigator, Chang Gung Memorial Hospital
Other Study IDs: 100-3793A3
Record Dates: First submitted 2017-08-22; First posted 2017-08-30 (Actual); Last update posted 2017-08-31 (Actual); Status verified 2017-08

CONDITIONS: Torticollis Congenital; Wryneck
Keywords: congenital muscular torticollis; wryneck; sternocleidomastoid; ultrasonography; digital analysis
MeSH Terms: conditions — Congenital torticollis; Torticollis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Wryneck: those with a condition

SUMMARY:
Torticollis is a clinical sign or symptom that could be the result of a variety of underlying disorders. Among the etiologies, Congenital muscular torticollis (CMT) with impairment of the sternocleidomastoid (SCM) is the most frequent cause of torticollis in infants. CMT is a postural deformity detected at birth or shortly after birth, primarily resulting from unilateral shortening and fibrosis of the SCM. Infants with CMT display head tilt to one side, which is often combined with rotation of the head to the opposite side. In 2002, Chih-Chin Hsu et al. reported that CMT could be classified into four types. The majority of Type I and II fibrosis improved after conservative treatment. However, Type III and Type IV had more probability in need of surgical correction. However, this categorization lacks of objective and quantitative measurement and can be different by subjective judgement of different physicians. The purpose of this study is tried to perform digital analysis of ultrasonography images to establish an objective, quantitative method and to assess its relevance with clinical symptoms and prognosis.

This study will collect the children younger than one year-old who were impressed or suspected to have torticollis in physical medicine and rehabilitation clinic to assess the relationship between digitalization results of ultrasound image and clinical manifestations and prognosis. Digital image analysis of ultrasound which contains both sides of the SCM in transverse and longitudinal view for comparison of lesion side and sound side will be performed after the initial enrollment and every six months later. Evaluation of clinical manifestations includes measurement of side difference of angles in bilateral neck lateral flexion, rotation and habitual head position will performed using an arthrodial protractor by a trained member at the beginning of physical therapy and one month later, then every 2-3 months. All cases will be followed for 1 and a half years. We expect to find some typical characteristics of CMT through digital analysis of the SCM. These characteristics include the muscle thickness and intensity of echogenicity in the region of interest. The Pearson's correlation will be performed to analyze the relevance of quantitative side differences in ultrasonography and clinical manifestations including side differences of neck rotation, lateral flexion and habitual head position between lesion sides and sound sides.

DETAILED DESCRIPTION:
Torticollis is a clinical sign or symptom that could be the result of a variety of underlying disorders. Among the etiologies, Congenital muscular torticollis (CMT) with impairment of the sternocleidomastoid (SCM) is the most frequent cause of torticollis in infants. CMT is a postural deformity detected at birth or shortly after birth, primarily resulting from unilateral shortening and fibrosis of the SCM muscle. Infants with CMT display head tilt to one side, which is often combined with rotation of the head to the opposite side. CMT is estimated to occur in one infant of every 300 live births. Plagiocephaly is reported as a coexisting impairment in 80% to 90.1% of children with CMT.

The pathophysiology and etiology of SCM impairment in CMT is still unknown. Prominent theories related to the cause of SCM impairment in CMT include intrauterine crowding, muscle trauma during a difficult delivery, soft tissue compression leading to compartment syndrome, and congenital abnormalities of soft tissue differentiation within the SCM muscle.

Children with CMT can be assigned to one of three clinical subgroups: 1) children with a palpable swelling or pseudotumor of the sternocleidomastoid, 2) children with SCM tightness but no tumor, and 3) children with all the features of muscular torticollis without muscle tightness or tumor.

In 2002, Chih-Chin Hsu et al. reported that CMT could be classified into four types. Type I denoted a heteroechoic mass in the affected muscles; Type II represented diffuse echogenic dots and lines against the hypoechoic background with no detectable mass. The alignment of perimysium appeared irregular instead of parallel on longitudinal sonograms; Type III indicated diffuse hyperechoic echogenicity along the entire muscle and almost no hypoechoic background could be seen; and Type IV had a hyperechoic band in the involved muscles. The study also evaluated the histology of each type of fibrosis. Type I and II fibrosis revealed hyperplastic fibrous tissue mingled with muscle fiber. Mature fibroblasts with complete absence of normal muscle tissue could be found in Type III fibrosis and the fibrotic bands in Type IV fibrosis. The majority of Type I and II fibrosis improved after conservative treatment. However, Type III and Type IV had more probability in need of surgical correction. However, this categorization lacks of objective and quantitative measurement and can be different by subjective judgement of different physicians. The purpose of this study is tried to perform digital analysis of ultrasonography images to establish an objective, quantitative method and to assess its relevance with clinical symptoms and prognosis.

General Design:

This study is planned to quantify ultrasonography image of wry neck patients by digital analysis.

Subjects:

This study will collect the children younger than 1 y/o who were impressed or suspected to have torticollis in physical medicine and rehabilitation clinic. The case number is estimated around 60 in a 3-year-period enrollment. . Exclusion criteria include torticollis by other known causes like strabismus, trauma, neurogenic problems, congenital malformation or bony deformity (e.g. hemivertebrae of cervical spine). Informed consent will be given to the parents before enrollment.

Investigation Steps:

1. Ultrasonography examination and digital analysis:

   Ultrasonography which contains both sides of the sternocleidomastoid muscle in transverse and longitudinal view for comparison of lesion side and sound side will be performed by expert physicians using a 14-megahertz linear-array transducer after the initial enrollment and every six months later. Digital analysis of the images will be carried by a member expert in computer science.
2. Evaluation of clinical manifestations:

   Evaluation of clinical manifestations includes measurement of side difference of angles in bilateral neck lateral flexion, rotation and habitual head position will performed using an arthrodial protractor by a trained member at the beginning of physical therapy and one month later, then every 2-3 months. Each measurement will be repeated 3 times to get the mean value. All cases will be followed for 1 and a half years, however, if the symptoms got completely recovery (the neck range of motion and position completely equal to sound side) or any complications resulting from the evaluation, the evaluation will be stopped.
3. Evaluation of influence of rehabilitation effect:

The parents will be inquired by a questionnaire one month later and then every 2-3 months to realize the treatment effect of the wry neck. The duration and frequency of massage and stretch programs by the therapist or the family or the other methods to treat the problem like wearing a neck collar, proper positioning… etc will be included in the semi-quantitative questionnaire.

Data Analysis:

Some representative image features will be expected to be computed from the SCM ultrasonic images. These features include area, both max and min Feret's diameters, and brightness of echogenicity in the region of interest. The ultrasonic image of the affected side would be compared with that of the sound side from their corresponding texture features. The Pearson's correlation will be performed to analyze the relevance of quantitative side differences of texture features in ultrasonography and clinical manifestations including side differences of neck rotation, lateral flexion and habitual head position between lesion sides and sound sides. Linear regression will be also used to adjust the influence of the treatment effect.

ELIGIBILITY:
Inclusion Criteria:

1. infants with congenital muscular torticollis and
2. age <12 months at diagnosis

Exclusion Criteria:

(1) wryneck caused by other known problems, including strabismus, trauma, neurogenic problems, congenital malformation, or bony deformity (e.g., hemivertebrae of the cervical spine)

Max Age: 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2013-04-30 (Actual); Primary Completion 2015-08-15 (Actual); Study Completion 2015-08-15 (Actual)

PRIMARY OUTCOMES:
cervical passive range of motion | From the date of beginning of physical therapy until the date of wryneck condition resolved or date of any complications resulting from the evaluation, whichever came first, assessed up to 18 months.
  Measurement with an arthrodial protractor by a trained physiotherapist at the beginning of physical therapy and one month later, then every 2-3 months. Each measurement will be repeated 3 times to get the mean value.. All cases will be followed for 1 and a half years, however, if the symptoms got completely recovery (the neck range of motion and position completely equal to sound side) or any complications resulting from the evaluation, the evaluation will be stopped.

SECONDARY OUTCOMES:
Area in cm^2 | From the date of initial enrollment until the date of wryneck condition resolved or date of any complications resulting from the evaluation, whichever came first, assessed up to 18 months.
  Ultrasonography which contains both sides of the sternocleidomastoid muscle in transverse and longitudinal view for comparison of lesion side and sound side will be performed by expert physicians using a 14-megahertz linear-array transducer after the initial enrollment and every six months later. Digital analysis of the images will be carried by a member expert in computer science. The area was measured in pixels on the original image. Thus, dividing by the pixels of one square centimeter on each sonogram, the unit of the area was converted to square centimeter.
Brightness of echogenicity in % | From the date of initial enrollment until the date of wryneck condition resolved or date of any complications resulting from the evaluation, whichever came first, assessed up to 18 months.
  Ultrasonography which contains both sides of the sternocleidomastoid muscle in transverse and longitudinal view for comparison of lesion side and sound side will be performed by expert physicians using a 14-megahertz linear-array transducer after the initial enrollment and every six months later. Digital analysis of the images will be carried by a member expert in computer science. The sonograms were grayscale images, and the mean gray value was measured from 0 to 255 in the image analysis software where zero was designated black and 255 was designated white. Therefore, the mean gray value was divided by 255 and then converted to a percentage. In this study, zero percent was designated black, and 100% was designated white and indicated the brightness of the echogenicity on the sonogram.
max Feret's diameter in cm | From the date of initial enrollment until the date of wryneck condition resolved or date of any complications resulting from the evaluation, whichever came first, assessed up to 18 months.
  Ultrasonography which contains both sides of the sternocleidomastoid muscle in transverse and longitudinal view for comparison of lesion side and sound side will be performed by expert physicians using a 14-megahertz linear-array transducer after the initial enrollment and every six months later. Digital analysis of the images will be carried by a member expert in computer science. The max Feret's diameter was measured in pixels on the original image. Thus, dividing by the pixels of one centimeter on each sonogram, the unit of the max Feret's diameter was converted to centimeter.
min Feret's diameter in cm | From the date of initial enrollment until the date of wryneck condition resolved or date of any complications resulting from the evaluation, whichever came first, assessed up to 18 months.
  Ultrasonography which contains both sides of the sternocleidomastoid muscle in transverse and longitudinal view for comparison of lesion side and sound side will be performed by expert physicians using a 14-megahertz linear-array transducer after the initial enrollment and every six months later. Digital analysis of the images will be carried by a member expert in computer science. The min Feret's diameter was measured in pixels on the original image. Thus, dividing by the pixels of one centimeter on each sonogram, the unit of the min Feret's diameter was converted to centimeter.

CONTACTS AND LOCATIONS:
Overall Officials: Chu-Hsu Lin, MD, Principal Investigator — Chang Gung Memorial Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cheng JC, Tang SP, Chen TM, Wong MW, Wong EM. The clinical presentation and outcome of treatment of congenital muscular torticollis in infants--a study of 1,086 cases. J Pediatr Surg. 2000 Jul;35(7):1091-6. doi: 10.1053/jpsu.2000.7833. PMID 10917303
- [Background] Canale ST, Griffin DW, Hubbard CN. Congenital muscular torticollis. A long-term follow-up. J Bone Joint Surg Am. 1982 Jul;64(6):810-6. PMID 7085709
- [Background] Hollier L, Kim J, Grayson BH, McCarthy JG. Congenital muscular torticollis and the associated craniofacial changes. Plast Reconstr Surg. 2000 Mar;105(3):827-35. doi: 10.1097/00006534-200003000-00001. No abstract available. PMID 10724239
- [Background] Cheng JC, Wong MW, Tang SP, Chen TM, Shum SL, Wong EM. Clinical determinants of the outcome of manual stretching in the treatment of congenital muscular torticollis in infants. A prospective study of eight hundred and twenty-one cases. J Bone Joint Surg Am. 2001 May;83(5):679-87. doi: 10.2106/00004623-200105000-00006. PMID 11379737
- [Background] Clarren SK, Smith DW, Hanson JW. Helmet treatment for plagiocephaly and congenital muscular torticollis. J Pediatr. 1979 Jan;94(1):43-6. doi: 10.1016/s0022-3476(79)80347-9. PMID 758420
- [Background] Cheng JC, Au AW. Infantile torticollis: a review of 624 cases. J Pediatr Orthop. 1994 Nov-Dec;14(6):802-8. PMID 7814599
- [Background] Dunn PM. Congenital postural deformities. Br Med Bull. 1976 Jan;32(1):71-6. doi: 10.1093/oxfordjournals.bmb.a071327. No abstract available. PMID 130955
- [Background] Ling CM, Low YS. Sternomastoid tumor and muscular torticollis. Clin Orthop Relat Res. 1972 Jul-Aug;86:144-50. doi: 10.1097/00003086-197207000-00020. No abstract available. PMID 5065412
- [Background] Davids JR, Wenger DR, Mubarak SJ. Congenital muscular torticollis: sequela of intrauterine or perinatal compartment syndrome. J Pediatr Orthop. 1993 Mar-Apr;13(2):141-7. PMID 8459000
- [Background] Tang S, Liu Z, Quan X, Qin J, Zhang D. Sternocleidomastoid pseudotumor of infants and congenital muscular torticollis: fine-structure research. J Pediatr Orthop. 1998 Mar-Apr;18(2):214-8. PMID 9531404
- [Background] Tang SF, Hsu KH, Wong AM, Hsu CC, Chang CH. Longitudinal followup study of ultrasonography in congenital muscular torticollis. Clin Orthop Relat Res. 2002 Oct;(403):179-85. doi: 10.1097/00003086-200210000-00026. PMID 12360024